CLINICAL TRIAL: NCT05407558
Title: Does the Menstrual Phase Affect Gastric Emptying? Prospective, Observational Study
Acronym: MAGUSG
Status: Completed | Type: Observational
Sponsor: Konya Meram State Hospital (Other)
Responsible Party: Principal Investigator, Betul Kozanhan, Ass.Prof., Konya Meram State Hospital
Other Study IDs: Menstrual Phase Gastric USG
Record Dates: First submitted 2022-05-27; First posted 2022-06-07 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-09

CONDITIONS: Gastric Contents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective observational study aimed to evaluate the relationship between menstrual phase cycles and gastric emptying in female volunteers of reproductive age.

DETAILED DESCRIPTION:
Volunteers included in the study will be evaluated for gastric emptying with USG in both phases of the menstrual phase. In each phase, volunteers will be evaluated for gastric emptying of both liquid food intake and a light meal. At first, 400 ml of water will be drunk after 10 hours of fasting, and gastric content will be evaluated with USG after 2 hours.

Secondly, after 10 hours of fasting, solid food intake will be evaluated. Then, after taking a light meal (toast and 200 ml tea), the volunteers will be evaluated by USG at the 6th hour.

ELIGIBILITY:
Inclusion Criteria:

* Female volunteers of reproductive age have had a regular menstrual cycle for at least six months

Exclusion Criteria:

* Pregnancy
* Stomach problem
* Using anticholinergics, opioids, and oral contraceptive drugs
* Hypothyroidism
* Diabetes mellitus
* Smokers

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — female volunteers with active menstrual cycles
Study Population: 24 healthy female volunteers who are of the reproductive age and have had a regular menstrual cycle for at least six
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2022-08-29 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
The difference in gastric volume between the two menstrual phases | 1 month
  gastric emptying with USG will be evaluated in both phases of the menstrual phase

CONTACTS AND LOCATIONS:
Locations (1):
- Betul Kozanhan, Konya, Turkey (Türkiye)